CLINICAL TRIAL: NCT03885453
Title: Construction of a Questionnaire on Panic Disorder and Agoraphobia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ulrike Willutzki (Other)
Responsible Party: Sponsor-Investigator, Ulrike Willutzki, Clinical Professor, University of Witten/Herdecke
Organization: University of Witten/Herdecke (Other)
Other Study IDs: 08/2018
Record Dates: First submitted 2018-12-05; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Panic Disorder; Panic Disorder With Agoraphobia; Agoraphobia; Agoraphobia With Panic Attacks; Depression
MeSH Terms: conditions — Panic Disorder; Agoraphobia; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Panic Disorder / Agoraphobia: Patients with Panic Disorder / Agoraphobia as major diagnosis
- Depression: Patients with Depression as major diagnosis

SUMMARY:
For the first time panic disorder and agoraphobia are included as separate disorders in the DSM-5. Thus, agoraphobia no longer represents a subcategory of panic disorder. To diagnose both of the disorders, questionnaires are the method of choice. However, there are no measuring instruments available free of charge in German-speaking countries. In order to improve this situation, the Witten Panic Disorder Questionnaire (WPF) and the Witten Agoraphobia Questionnaire (WAF) are constructed in accordance with the DSM-5 criteria. Both measuring instruments are included as a part of a ten instrument battery. WAF and WPF will be delivered to a patient sample of patients with panic disorder and/or agoraphobia as well as depressed patients (discriminant validity). Factor analyzes and item analyses will be conducted.

ELIGIBILITY:
Inclusion Criteria:

Panic Disorder / Agoraphobia / Depression diagnosis via diagnostic interview

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Panic Disorder / Agoraphobia / Depression
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Wittener Panik Fragebogen (WPF) | 5 min
  Self developed panic disorder questionnaire. Measures panic symptoms on one scale. Items are averaged. Range: 1-5. Higher values represent a worse outcome.
WAF | 10 min
  Self developed agoraphobia questionnaire. Measures agoraphobia symptoms on two scales (Fear and Avoidance). Items are averaged to calculate the subscales. Range: 1-5 (Fear); 1-3 (Avoidance). Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Agoraphobic Cognition Questionnaire (ACQ) | 5 min
  Chambless et al. (1985); Ehlers et al. (1993). The questionnaire measures anxious thoughts on two scales: Loss of Control and Physical Concerns. Items are averaged to calculate the subscales. Range: 1-5. A total score is calculated by averaging all items. Higher values represent a worse outcome.
Body Sensations Questionnaire (BSQ) | 5 min
  Chambless et al. (1985); Ehlers et al. (1993). The questionnaire measures body sensations that may occur in a feared situation. Items are averaged to calculate a total score. Range: 1-5. Higher values represent a worse outcome.
Mobility Inventory (MI) | 10 min
  Chambless et al. (1985); Ehlers et al. (1993). The questionnaire measures avoidance of agoraphobic situations on two scales (Avoidance Alone and Avoidance Accompanied). Items are averaged to calculate the scales. Range: 1-5. Higher values represent a worse outcome.
Agoraphobic Self-Statements Questionnaire (ASQ) | 5 min
  Hout et al. (2001). Measures agoraphobic statements on two scales (positive self-statements and negative self-statements). Items are averaged. Range: 0-4. Higher values represent a better outcome on the positive scale and a worse outcome on the negative scale.
Agoraphobic Cognitions Scale - extended version (ACS+) | 5 min
  Hoffart et al. (1992). Measures fearful cognitions on three scales (fear of bodily incapacitation, fear of losing control, and fear of acting embarrassingly). Items are averaged to calculate the scales. Range: 0-4. Higher values represent a worse outcome.
Patient Health Questionnaire - D (PHQ-D) - Subscale Panic Syndrome | 5 min
  Spitzer, Kroenke & Williams (1999); Löwe et al. (2002). The questionnaire measures symptoms on modular scales. The panic syndrome subscale is calculated by summing up all 11 items. The scale ranges from 0 to 1. The sum score ranges from 0 to 11. Higher values represent a worse outcome.
Brief Symptom Inventory (BSI) | 10 min
  Derogatis & Melisaratos (1983); Franke (2000). Measures psychopathological symptoms on nine scales (Somatization, Obsessive-Compulsive, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, Psychoticism). Items are averaged to calculate the subscale scores. Range: 0-4. The Global Severity Index (GSI) is calculated by averaging all items. Higher values represent a worse outcome.
Beck Depression Inventory (BDI) | 10 min
  Beck et al. (1961). Measures depressive symptoms on one scale. Items summed up to calculate the toal score. The scale ranges from 0 to 3. The sum score ranges from 0 to 63. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Witten/Herdecke University, Witten, North Rhine-Westphalia, Germany